CLINICAL TRIAL: NCT04922151
Title: A Randomized, Double Masked, Multicenter, Phase II Study Assessing the Safety and Efficacy of 601 Versus Ranibizumab in Patients With Visual Impairment Due to Pathological Myopic Choroidal Neovascularization (pmCNV)
Brief Title: 601 Versus Ranibizumab in Patients With Pathological Myopic Choroidal Neovascularization (pmCNV)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SSGJ-601-pmCNV-II-01
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Pathological Myopic Choroidal Neovascularization
Keywords: VEGF; pmCNV; antibody
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group I (Experimental): 601 1.25mg
  Interventions: Drug: 601
- group II (Active Comparator): Ranibizuman 0.5 mg
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: 601 — intravitreal recombinant humanized anti-VEGF monoclonal antibody
  Arms: group I
Drug: Ranibizumab — intravitreal recombinant humanized anti-VEGF monoclonal antibody
  Arms: group II

SUMMARY:
To evaluate the safety and efficacy of intravitreal recombinant humanized anti-VEGF monoclonal antibody in patients with visual impairment due to pmCNV

DETAILED DESCRIPTION:
Following a 14-day maximum screening period, patients will be randomized and followed for approximately 36 weeks. Treatment visits will be scheduled in 4-week intervals. After 1 initial injection of 601 or ranibizumab (loading phase), subjects will enter an individualized flexible treatment (IFT) phase (week 4 to week 32). During the IFT phase, an assessment of disease stability will be performed at each monthly visit and subjects will receive either an injection or not. Safety and efficacy outcomes will continue to be evaluated up to a period of 36 weeks unless the patient is withdrawn or discontinues the study.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent form and willing to be visited at the time specified in the trial
* Male or Female, at least 18 years of age
* The study eye must meet the following criteria
* Diagnosed with active choroidal neovascularization secondary to pathological myopia
* BCVA score between 78 and 24 letters, inclusive, using ETDRS visual acuity testing charts (approximate Snellen equivalent of 20/32 to 20/320)
* No optometric media opacity and pupil abnormal
* BCVA score ≥ 34 letters in the fellow eye, using ETDRS visual acuity testing charts (approximate Snellen equivalent of 20/200)

Exclusion Criteria:

* CNV secondary to other causes (except pathological myopia), such as neovascularage-related macular degeneration (nAMD), polypoid choroidal vascular disease (PCV), and secondary injury
* The fovea has fibrosis and organochemical foci or scar or atrophy that obviously involves the fovea and causes irreversible vision loss;
* Previous use of intraocular or periocular steroids within 3 months prior to baseline, or previous use of dexamethasone intravitreal implant within 6 months prior to enrollment;
* PDT, Macular laser photocoagulation (focal/grid), vitrectomy or keratoplasty in the study eye at any time prior to baseline. Panretinal laser photocoagulation，YAG laser treatment or any other ocular surgeries (e.g. cataract surgery ) in the study eye within 3 months prior to the baseline
* Aphakia (except IOL) or posterior capsular defect (except YAG posterior capsulotomy after intraocular lens implantation surgery)

For Any Eye:

* Any eye has active ocular infections (e.g. blepharitis, conjunctivitis, keratitis, scleritis, uveitis, endophthalmitis)
* History of intravitreal use of anti-VEGF drugs (e.g. ranibizumab，bevacizumab，aflibercept, conbercept, etc.) in any eye within 3 months prior to baseline

General Exclusion Criteria:

* History of allergy to fluorescein sodium and allergies to protein products for treatment or diagnosis
* History of stroke (cerebrovascular accident), myocardial infarction, active disseminated intravascular coagulation or pronounced bleeding tendency in the past 6 months prior to baseline
* Diagnosed systemic immune diseases (e.g. ankylosing spondylitis, systemic lupus erythematosus, Behcet's disease, rheumatoid arthritis, scleroderma etc.)
* any uncontrolled clinical problem (e.g. AIDS, active hepatitis, serious mental, neurological, cardiovascular, respiratory and other systemic diseases or malignant tumors, etc.). Malignant tumors with no metastasis or recurrence within 5 years or cancers in situ cancers are not excluded.
* History of system use of anti-VEGF drugs (e.g. bevacizumab) within 3 months prior to baseline

Laboratory Exclusion Criteria:

* Liver dysfunction (ALT or AST is 2 times higher than the upper limit of normal value in the local laboratory). Renal function impairment (Cr is 1.5 times higher than the upper limit of normal values in the local laboratory)
* Abnormal coagulation function (prothrombin time >= the upper limit of normal value for 3 seconds) and activated partial thromboplastin time >= the upper limit of normal value for 10 seconds);

Other Exclusion Criteria:

* Non-use of effective contraception during childbearing age (except for women with spontaneous admonishment of more than 12 months)
* Pregnancy and lactation women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-04 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in best-corrected visual acuity (BCVA) at Week 12 | Baseline to Week 12
  Assessed with ETDRS visual acuity testing charts.

SECONDARY OUTCOMES:
Average Change of BCVA on each visit compared to baseline. | Baseline to Week 36
  Assessed with ETDRS visual acuity testing charts.
Change from baseline in central retina thickness (CRT) on each visit | Baseline to Week 36
  OCT (optical coherence tomography) was used to assess central retina thickness (CRT) representing the average retinal thickness of the central 1 mm diameter subfield around the foveal center.
Proportion of study eyes with a gain ≥ 5, 10 and 15 letters in BCVA on each visit compared to baseline | Baseline to Week 36
  Assessed with ETDRS visual acuity testing charts.
Number of injections from Week 4 to Week 36 | Week 4 to Week 36
  Number of administered injections
Incidence of ocular and non-ocular AEs up to Week 36 | Baseline to Week 36
  Incidence of ocular and non-ocular AEs
Blood concentrations of 601 | Baseline, Week 4, Week 12, Week 24 and Week 36.
  Steady-state blood concentrations of 601
Blood concentrations of VEGF | Baseline, Week 4, Week 12, Week 24 and Week 36.
  Detection of VEGF blood concentration
Immunogenicity of 601 | Baseline, Week 4, Week 12, Week 24 and Week 36.
  Detection of blood Anti-drug antibody (ADA) status. If ADA was positive, Neutralization antibody (Nab) will be tested

CONTACTS AND LOCATIONS:
Overall Officials: YouXin Chen, PHD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No